CLINICAL TRIAL: NCT04644757
Title: Feasibility and Efficacy of Remotely Monitored Home-based Listening to Preferred Music for Pain in Older Adults With Low Back Pain: A Pilot Study of Feasibility and Acceptability
Brief Title: Feasibility and Efficacy of Remotely Monitored Home-based Listening to Preferred Music for Pain in Older Adults With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Martel Scholarship (Unknown)
Responsible Party: Principal Investigator, Setor K. Sorkpor, Student, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-20-1092
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Other: Music Listening

INTERVENTIONS:
Other: Music Listening — The study will employ an individual receptive relaxation music method with participants selecting music based on their preference from a selection of various styles from the MUSIC CARE© app. The music intervention will last 20 minutes per session and will be administered twice daily for 4 consecutive days. Participants will be given an electronic tablet with the MUSIC CARE© app loaded on it and trained on how to access the app to select their preferred style of music.Participants will be instructed to use the provided headphone during all interventions and to sit in a quiet area while wearing an ocular mask to avoid distractions.The PI will remotely monitor each of the music intervention sessions in real-time monitoring via a secured video conferencing interface to ensure adherence to study protocol.

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of listening to 20 minutes of preferred style of music twice-daily for 4 consecutive days on pain among 20 community-dwelling older adults with lower back pain (LBP)

ELIGIBILITY:
Inclusion Criteria:

* self-report of Lower back pain (LBP)
* LBP in the past 3 months with an average rating of at least 30 on a 0 - 100 NRS for pain
* intact cognition
* no plans to change their pain medication regimens during the study time
* can read and understand English
* can travel to the study center
* agree to sign an informed consent

Exclusion Criteria:

* deaf or have severe hearing loss
* pregnant or lactating
* have an implantable pain-reducing device
* history of hospitalization within the preceding year for psychiatric illness
* diagnosis of Raynaud's disease
* have a functional limitation that requires the use of an ambulatory aid such as a cane, walker, or wheelchair
* history of brain surgery, brain tumor, or stroke
* severe depression (PROMIS Depression T-score ≥ 70) (Kroenke et al., 2020)
* severe anxiety (PROMIS Anxiety ≥ 70) (American Psychiatric Association, 2013)
* Mini-Mental State Examination score less than 24 (Creavin, Wisniewski, Noel-Storr, et al., 2016)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Enrollment rate: Assessed as number enrolled or number who met inclusion criteria | 6 months from start of study
Attrition rate | 6 months from start of study
  Assessed as number not completing the study divided by number enrolled at baseline
Adherence rate | 6 months from start of study
  Assessed as number completing all measures divided by number enrolled
Treatment acceptability: Measured by the treatment acceptability and preference scale(TAP | Baseline
  Assess perceived acceptability of treatment using TAP in four categories of appropriateness, effectiveness, suitability, and willingness to adhere on a scale ranging from 0 (not at all) to 4 (very much).
Treatment acceptability: Measured by the treatment acceptability and preference scale(TAP) | 5 days after baseline(1 day after completion of intervention)
  Assess perceived acceptability of treatment using TAP in four categories of appropriateness, effectiveness, suitability, and willingness to adhere on a scale ranging from 0 (not at all) to 4 (very much).

SECONDARY OUTCOMES:
Pain as measured by the numerical rating scale (NRS) | Baseline
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 7 days will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Pain as measured by the numerical rating scale (NRS) | day 1
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 24 hours will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Pain as measured by the numerical rating scale (NRS) | day 2
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 24 hours will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Pain as measured by the numerical rating scale (NRS) | day 3
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 24 hours will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Pain as measured by the numerical rating scale (NRS) | day 4
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 24 hours will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Pain as measured by the numerical rating scale (NRS) | post intervention (day 5)
  Self-reported mean clinical pain intensity defined as the average pain intensity experienced in the past 24 hours will be measured using the 101-point NRS where 0 means no pain and 100 means worst imaginable pain.
Anxiety as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form | Baseline
  The PROMIS Anxiety Short Form has 8 items with each item on the measure being rated on a 5-point scale (1-5) , a higher number indicating a worse outcome
Depression as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form | Baseline
  The PROMIS Depression Short Form has 8 items with each item on the measure being rated on a 5-point scale (1-5) , a higher number indicating a worse outcome
Change in brain activation in the motor and somatosensory cortex as measured by functional near-infrared spectroscopy (fNIRS) | Baseline and post-intervention (Day 5)
  Pain-related measure of hemodynamic response function will be measured during pressure pain stimulation using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) with three semiconductor lasers at 780, 805, and 830 nm.
Change in conditioned pain modulation (CPM) | Baseline and post-intervention (Day 5)
  Conditioned pain modulation will measure the difference in pressure pain threshold before and after a painful "conditioning stimulus" is applied to test central pain inhibition. The conditioning stimulus will involve the immersion of one hand in a cold-water bath. The pressure pain tolerance will be evaluated following a conditioning stimulus condition
Change in heart rate variability (HRV) | Baseline and post-intervention (Day 5)
  Heart rate variability will be assessed as an indicates the sympathetic nervous system status using lead II arrangement with an MP160 Data Acquisition Systems (Biopac Systems, Inc., Goleta, CA, U.S.A.).

CONTACTS AND LOCATIONS:
Overall Officials: Setor K Sorkpor, MPH,MSN,RN-BC, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No